CLINICAL TRIAL: NCT06047093
Title: Evaluation of the Intrahepatic Hepatitis B Virus Reservoir and Its Immunological Characteristics in Chronically HBV-infected Patients - Pilot Study
Brief Title: Fine Needle Aspiration (FNA) Evaluation of the Intrahepatic HBV Reservoir and Its Immunological Characteristics in Chronically HBV-infected Patients
Acronym: RES-HBV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL23_0275
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Chronic Hepatitis b
Keywords: Hepatitis B; HBV; cccDNA; functional cure; FNA; HBsAg
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Five groups according to HBsAg quantification (3 distinct groups with or without nucleoside analogues), HDV co-infection and HBsAg loss.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- HBsAg <100 IU/ml (Experimental): Patients chronically mono-infected with HBV, whose HBsAg is less than 100 IU/ml (patients treated or not with NA)
  Interventions: Procedure: Investigation of the intrahepatic compartment using the fine needle aspiration (FNA) technique; Biological: Creation of a serum biobank; Other: FNA feasibility and acceptability questionnaire
- HBsAg between 100 and 3000 IU/ml (Experimental): Patients chronically mono-infected with HBV, with HBsAg levels >100 and <3000 IU/ml (patients treated or not with NA).
  Interventions: Procedure: Investigation of the intrahepatic compartment using the fine needle aspiration (FNA) technique; Biological: Creation of a serum biobank; Other: FNA feasibility and acceptability questionnaire
- HBsAg ≥ 3000 IU/ml (Experimental): Patients chronically mono-infected with HBV, with HBsAg levels ≥ 3000 IU/ml (patients treated or not with NA).
  Interventions: Procedure: Investigation of the intrahepatic compartment using the fine needle aspiration (FNA) technique; Biological: Creation of a serum biobank; Other: FNA feasibility and acceptability questionnaire
- Loss of HBsAg (spontaneously or under NA) (Experimental): Patients with loss of HBsAg (spontaneously or under NA). This group will allow comparison of the HBsAg loss immuno-virological profile with that of patients with active infection and varying levels of HBsAg (groups 1-3 and 5) and aid in identifying of predictors of functional cure. The identification of determinants of HBV functional cure is fundamental and is comparable to investigations that have been carried out in HIV-infected "elite controllers".
  Interventions: Procedure: Investigation of the intrahepatic compartment using the fine needle aspiration (FNA) technique; Biological: Creation of a serum biobank; Other: FNA feasibility and acceptability questionnaire
- Patients co-infected with HBV and HDV (Experimental): Patients co-infected with HDV (positive HDV viral load), regardless of HBsAg level (presence or absence of HBV or HDV treatment)
  Interventions: Procedure: Investigation of the intrahepatic compartment using the fine needle aspiration (FNA) technique; Biological: Creation of a serum biobank; Other: FNA feasibility and acceptability questionnaire

INTERVENTIONS:
Procedure: Investigation of the intrahepatic compartment using the fine needle aspiration (FNA) technique — The FNA will be performed at the Croix Rousse digestive pathology day hospital of the Hospices Civils de Lyon by a doctor from the hepatology department who has been trained to perform FNA.
  After echography, a subcutaneous anesthesia with LIDOCAÏNE is administered. Two FNA passages will be performed for virological and immunological analyses. The patient will be monitored in the supine position for 1 hour after the procedure.
  A single FNA will be performed during the study.
Biological: Creation of a serum biobank — 42ml blood sample for study of circulating peripheral blood mononuclear cells (PBMC) and new circulating hepatitis B markers. These samples will enable us to gain a better understanding of peripheral immune responses and to correlate intrahepatic virological data with new serum markers of HBV.
Other: FNA feasibility and acceptability questionnaire — An FNA feasibility and acceptability questionnaire carried out at inclusion (V1) and after the FNA has been performed.

SUMMARY:
Two hundred and ninety-six million people worldwide are chronically infected with the hepatitis B virus (HBV), with around 750,000 deaths each year linked to the development of cirrhosis or hepatocellular carcinoma. Current treatments based on nucleoside analogues (NA) achieve virological cure in only 5% of cases at 10 years. The virological persistence of HBV is explained by the persistence of cccDNA (covalently-closed circular DNA) in the nucleus of hepatocytes. Complex and poorly understood interactions between immunological and virological responses explain the persistence of ccccDNA. A better understanding of the immunological and virological interactions of the intrahepatic compartment during chronic HBV infection is needed to better understand the mechanisms of viral persistence and for research and development of new drugs to achieve the goal of a functional cure for HBV (defined as the prolonged loss of Hepatitis B surface antigen (HBsAg) after cessation of treatment, associated with a decrease in intrahepatic cccDNA or its transcriptional inactivation).

The intra-hepatic compartment can be explored by liver biopsy. A fine needle aspiration (FNA) technique is used to characterize primary hepatic tumors, with fewer complications than liver biopsy. One study has validated its use for immunological exploration of the intra-hepatic compartment. Finally, a recently published study confirms a correlation between FNA and liver biopsy virological markers in patients with chronic HBV infection. However, no combined immuno-virological study has been carried out to explore this intra-hepatic compartment by FNA in patients with chronic HBV infection.

The investigators will assess the intrahepatic compartment of patients chronically infected with HBV (+/- hepatitis Delta (HDV)) to understand the mechanisms of viral persistence and characterize host immune responses to HBV. These investigations will make it possible to determine the immuno-virological profiles of patients who would benefit from intensification of antiviral treatment or, potentially, discontinuation of antiviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years of age)
* Patients chronically infected with hepatitis B virus at any stage of infection
* Nucleoside Analogues-treated or untreated
* Co-infected or not with HDV
* Included in the prospective CirB-RNA study (part of the CirB-RNA university research program) (ID-RCB : 2018-A02558-47, NCT03825458)
* Patient informed of the study and having signed a consent form

Exclusion Criteria:

* Pregnant, parturient or breast-feeding women,
* Patients with decompensated cirrhosis
* Patients with hepatocellular carcinoma (suspected or proven),
* Liver transplant patients (even if liver transplantation for HBV),
* Patients co-infected with HCV (positive serum viral load) and/or HIV (regardless of serum viral load).
* Patients participating at the time of inclusion in an interventional study
* Persons under psychiatric care,
* Persons admitted to a health or social institution for purposes other than research
* Adults under legal protection (legal guardianship, tutorship, curatorship)
* Persons not affiliated to a social security scheme or beneficiaries of a similar scheme.
* Patients with abdominal skin lesions and/or infections.
* Contraindication to lidocaine administration (allergy or hypersensitivity to the product).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2028-03-08 (Estimated); Study Completion 2028-03-08 (Estimated)

PRIMARY OUTCOMES:
Interaction between immune response against HBV and intrahepatic HBV viral load | Baseline
  The main objective is to analyze the interaction between intrahepatic adaptive immune responses (Number and functional profile of CD4+ T lymphocytes and CD8+ B lymphocytes) and intrahepatic HBV viral load obtained from FNA.
  Immune and virological responses obtained from the FNA performed.

SECONDARY OUTCOMES:
Correlation between intrahepatic HBV markers and HBV serum markers | Baseline, 6 months, 12 months, 18 months and 24 months after inclusion
  Correlate intrahepatic markers of HBV (copies of intra-hepatic HBV, cccDNA, cccDNA transcriptional activity, HBV RNA) and new serum markers of HBV cure (circulating viral RNA, HBcrAg) and their evolution over time Intrahepatic HBV markers obtained from the FNA performed. New serum markers are taken at each visit for 24 months
Intrahepatic immune and virological responses in relation to the phases of HBV or HDV co-infection | Baseline
  Analyze immune (copies of intra-hepatic HBV, cccDNA and cccDNA transcriptional activity) and virological responses (Number and functional profile of CD4+ T lymphocytes and CD8+ B lymphocytes) as a function of the phases of chronic HBV infection and co-infection with HDV.
  Immune and virological responses obtained from the FNA performed.
Intrahepatic immunological and virological responses according to the presence or absence of NA | Baseline
  Analyze immune (copies of intra-hepatic HBV, cccDNA and cccDNA transcriptional activity) and virological responses (Number and functional profile of CD4+ T lymphocytes and CD8+ B lymphocytes) according to the presence or absence of NA treatment.
  Immune and virological responses obtained from the FNA performed.
Assessing patient tolerance and acceptability of FNA | Baseline (before then after FNA)
  A questionnaire on the acceptability and tolerance of FNA will be given to each patient at the inclusion visit and after FNA has been performed (15-30 days after inclusion).
  An FNA feasibility and acceptability questionnaire carried out at inclusion (V1) and after FNA had been performed.

CONTACTS AND LOCATIONS:
Overall Officials: Fabien ZOULIM, PU-PH, Principal Investigator — Service d'Hépatologie de l'Hopital Croix-Rousse
Locations (1):
- Hepatology Department - Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No